CLINICAL TRIAL: NCT05970250
Title: Effect Of Whole Body Vibration Versus Weight Bearing Exercises On Osteoporosis In Breast Cancer Patients After Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mahrous Abdel-Hamed Ahmed Elgendy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Eman Mahrous Abdel-Hamed Ahmed
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Osteoporosis; Breast Cancer
MeSH Terms: conditions — Osteoporosis; Breast Neoplasms | interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole body vibration group (Experimental): In this group (the first study group) fifteen breast cancer patients after receiving chemotherapy within 3-6 months and complaining from osteoporosis were received the whole body vibration, 20 minutes 3 times per week for 2 months and drug therapy (vitamin D supplements and calcium).
  Interventions: Other: Whole body vibration group; Drug: vitamin D supplements and calcium
- Weight bearing exercises group (Experimental): In this group (the second study group) fifteen breast cancer patients after receiving chemotherapy within 3-6 months and complaining from osteoporosis were received aerobic exercise on treadmill as form of weight bearing exercise 20 minutes 3 times per week for 2 months and drug therapy (vitamin D supplements and calcium).
  Interventions: Other: Weight bearing exercises; Drug: vitamin D supplements and calcium
- drug therapy group (Other): In this group (control group) fifteen breast cancer patients after receiving chemotherapy within 3-6 months and complaining from osteoporosis were received only drug therapy (vitamin D supplements and calcium. Measurements were conducted before starting the treatment as a first record, at end of the second month of treatment as second record and make follow up after 3 months as final record.
  Interventions: Drug: vitamin D supplements and calcium

INTERVENTIONS:
Other: Whole body vibration group — Whole body vibration apparatus (model Power plate -my5tm, made in United States) with frequency 30 - 40 Hz was used for the whole body vibration program by reciprocating vertical displacements on the left and right side of a fulcrum.
  Arms: Whole body vibration group
Other: Weight bearing exercises — Electronic treadmill Kettler- marathon model No 7899-800, made in Germany (as form of weight bearing exercises), which was adjusted to the subject's comfortable walking speed. Generally, during the treadmill training, its speed and inclination are electronically adjusted, and it is also provided with a control panel to display the exercise parameters. It allows for the comfortable running without joint or back pains through a perfect combination between aluminium-pertinax running deck, shock absorbers and overall shock-damping design.
  Arms: Weight bearing exercises group
Drug: vitamin D supplements and calcium — vitamin D supplements and calcium

SUMMARY:
Chemotherapy can damage bone marrow and therefore impair the production of white blood cells, platelets and red blood cells with the resulting anemia and osteoporosis.

DETAILED DESCRIPTION:
Purposes of this study were:

1. To determine the therapeutic efficacy of the whole-body vibration (WBV) in improving osteoporosis in breast cancer patients after receiving chemotherapy within 3-6 months.
2. To determine the therapeutic efficacy of the weight bearing exercise in improving osteoporosis in breast cancer patients after receiving chemotherapy within 3-6 months.
3. To gain knowledge about the whole-body vibration (WBV) and the weight bearing exercise in improving osteoporosis in breast cancer patients after receiving chemotherapy within 3-6 months.
4. To share in designing an ideal protocol for the treatment of the osteoporosis in breast cancer patients after receiving chemotherapy within 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients after receiving chemotherapy within 3-6 months and complaining from osteoporosis.
* Their age ranges from 35-55 years old.
* All patients will have the same medical and nursing care.
* All the patients will receive a good explanation of treatment and measurement device.
* They are neurologically free.

Exclusion Criteria:

Patients will be excluded from this study for any of the following causes:

* Uncooperative patients.
* Instability of patient's medical condition.
* Association of another medical problem.
* Patients who have diabetes.
* Patients who have history of medical chronic relevant diseases.
* Patients who have acute or chronic hepatitis.
* Patients who have pacemaker.
* Patients who have genitourinary infections.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Assessing the change in bone mineral density | at baseline and after 2 months of intervention
  By using DEXA (dual-energy X-ray absorptiometry): Dual-energy X-ray absorptiometry (DEXA) is a clinically proven method of measuring bone mineral density (BMD) in the lumbar spine, proximal femur, forearm, and whole body. It is used primarily in the diagnosis and management of osteoporosis and other disease states characterized by abnormal BMD, as well as to monitor response to therapy for these conditions .

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elgendy, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided